CLINICAL TRIAL: NCT06807749
Title: PrEmenopausal bReaSt cancEr adjuVant thERapy Benefit According to OncotypE DX Test
Brief Title: Adjuvant Treatment in Premenopausal Breast Cancer
Acronym: PERSEVEREX
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Collaborators: Clinical Research Technology S.r.l. (Industry)
Responsible Party: Sponsor
Other Study IDs: 7296
Record Dates: First submitted 2025-01-10; First posted 2025-02-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)
Keywords: Premenopausal early breast cancer; Oncotype Dx

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- node negative (pN0): Patients with node negative (pN0) diagnosis and availability of Recurrence Score at Oncotype Dx test
- node positive (pN1): Patients with node positive (pN1) diagnosis and availability of Recurrence Score at Oncotype Dx test

SUMMARY:
Multicentric retroprospective observational study to collect outcome in premenopausal breast cancer patients who undergone the 21-multigene assay Oncotype DX from 1st January 2013 to 31st December 2022 and adjuvant treatment.

DETAILED DESCRIPTION:
Premenopausal patients who undergone the 21-multigene assay Oncotype DX from 1st January 2013 to 31st December 2022 with any Recurrence Score (RS) and pathological nodal status pN0/pN1 will be included in the study. The study will collect clinical-pathological, genomic characteristics, adjuvant treatments (chemotherapy, endocrine therapy with/without OFS), and survival outcome (iDFS).

ELIGIBILITY:
Inclusion Criteria:

1. Female, premenopausal and ≥18 years age patients.
2. Agree to participate in study and signing informed consent or declaration in lieu of informed consent form, if applicable
3. Histological diagnosis of early breast cancer hormone positive (ER and/or PgR), HER2-negative.
4. Pathological nodal stage of pN0 or pN1 (1-3 nodes) and pathological tumor stage of pT1 to pT3.
5. Surgery for primary breast cancer and axillary staging by sentinel node biopsy or axillary lymph node dissection (ALND).
6. Availability of 21-multigene assay Oncotype DX recurrence score results performed according to physician choice from 1st January 2013 to 31st December 2022
7. Availability of clinical and pathological information.
8. Availability of information about adjuvant treatment received.
9. Availability of patient' outcome information (relapse, site of relapse, survival).

Exclusion Criteria:

1. Evidence of distant metastases
2. Inflammatory breast cancer
3. Neoadjuvant treatment
4. No surgery for primary breast cancer and axillary staging
5. Patients not tested with 21-multigene assay Oncotype DX

Max Age: 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Female
Study Population: Patients with premenopausal early breast cancer HR+ HER2 negative diagnosis with any Recurrence Score (RS) and pathological nodal status pN0/pN1 and who underwent the 21-multigene assay Oncotype DX from 1st January 2013 to 31st December 2022 and adjuvant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease-Free Survival (iDFS) at 5 years | up to 30 months
  The primary endpoint of the study will be the invasive Disease-Free Survival (iDFS) at 5 years among pN0 and pN1 premenopausal breast cancer patients in subgroups formed according to their genomic risk according to 21- multigene assay Oncotype DX.

SECONDARY OUTCOMES:
To describe the effect of the different adjuvant treatments according to clinical and genomic risk | up to 30 months
  Descriptive statistics, statistical measure of association, and logistic binomial regression modeling of the association measures between the iDFS at 5 years and explicative variables including adjuvant treatment received (chemo/endocrine therapy; endocrine therapy with or without OSF), pathological tumor status, and genomic risk score according to 21-multigene assay Oncotype DX.

CONTACTS AND LOCATIONS:
Overall Officials: Antonella Palazzo, Principal Investigator — Fondazione Policlinico Gemelli, IRCCS; Alessandra Fabi, Study Chair — Fondazione Policlinico Gemelli, IRCCS
Locations (1):
- Clinical Research Technology, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No